CLINICAL TRIAL: NCT01489020
Title: Multicentre Phase I Randomized Double Blind Placebo Controlled Study of Subcutaneous Immunotherapy in Subjects With Allergic Rhinoconjunctivitis ± Asthma Sensitised to Dermatophagoides Pteronyssinus.
Brief Title: Subcutaneous Immunotherapy in Patients Sensitized to Dermatophagoides Pteronyssinus (DPT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-DPT-P1-001; 2009-016277-15 (EudraCT Number)
Record Dates: First submitted 2011-12-02; First posted 2011-12-09 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-01

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergy; Immunotherapy; Allergic Rhinoconjunctivitis; D. pteronyssinus; house dust allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A active (Experimental): 6 administrations and 5 weeks duration
  1. Vial 2: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals
  2. Vial 3: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals.
  Interventions: Biological: subcutaneous immunotherapy with DPT extract
- Group A placebo (Placebo Comparator): 6 administrations and 5 weeks duration
  1. Vial 2: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals
  2. Vial 3: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals.
  Interventions: Biological: Subcutaneous depot placebo
- group B active (Experimental): 8 administrations and 7 weeks duration
  1. Vial 1: 0.2 ml at 1 week intervals
  2. Vial 2: 0.1 ml, 0.2 ml, 0.4 ml at 1 week intervals
  3. Vial 3: 0.1 ml, 0.2 ml, 0.4 ml and 0.5 ml at 1 week intervals
  Interventions: Biological: subcutaneous immunotherapy with DPT extract
- Group B placebo (Placebo Comparator): 8 administrations and 7 weeks duration
  1. Vial 1: 0.2 ml at 1 week intervals
  2. Vial 2: 0.1 ml, 0.2 ml, 0.4 ml at 1 week intervals
  3. Vial 3: 0.1 ml, 0.2 ml, 0.4 ml and 0.5 ml at 1 week intervals
  Interventions: Biological: Subcutaneous depot placebo
- Group C active (Experimental): 8 administrations, 2 administrations in the same day. 1 week interval between 2 doses, during 3 weeks.
  1. Week 1: vial 2 - 2 administrations of 0.1 ml with 30 minute interval
  2. Week 2: vial 2 - 0.2 ml and 0.3 ml with 30 minute interval
  3. Week 3: vial 3 - 2 doses of 0.1 ml with 30 minute interval
  4. Week 4: vial 3 - 0.2 ml and 0.3 ml with 30 minute interval
  Interventions: Biological: subcutaneous immunotherapy with DPT extract
- Group C placebo (Placebo Comparator): 8 administrations, 2 administrations in the same day. 1 week interval between 2 doses, during 3 weeks.
  1. Week 1: vial 2 - 2 administrations of 0.1 ml with 30 minute interval
  2. Week 2: vial 2 - 0.2 ml and 0.3 ml with 30 minute interval
  3. Week 3: vial 3 - 2 dose of 0.1 ml with 30 minute interval
  4. Week 4: vial 3 - 0.2 ml and 0.3 ml with 30 minute interval
  Interventions: Biological: Subcutaneous depot placebo

INTERVENTIONS:
Biological: subcutaneous immunotherapy with DPT extract — Increasing doses of subcutaneous immunotherapy in three different scales up to the maximum dose of 500 TSU (Treatment Standardized Units)
  Other Names: DPT depot vaccine
  Arms: Group A active; Group C active; group B active
Biological: Subcutaneous depot placebo — Increasing doses of subcutaneous depot placebo in three different scales
  Arms: Group A placebo; Group B placebo; Group C placebo

SUMMARY:
Based on EMA (European Medicines Agency) new guidelines on the clinical development of products for immunotherapy for the treatment of allergic diseases the aim of this study was to assess safety and tolerability of 3 different subcutaneous immunotherapy dose escalations in patients allergic to Dermatophagoides pteronyssinus.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with allergic rhinoconjunctivitis with or without asthma against DPT during a minimum of 1 year prior to study participation.
2. Patients must sign the informed consent form.
3. Patients must be between 18 and 60 years of age.
4. Patients who obtained a prick test result greater or equal to 3 mm diameter and a specific IgE greater or equal to class 2 (CAP/PHADIA) to DPT.
5. Patients will preferably be monosensitized to DPT. In the case of polysensitized patients they can only be included if other sensitizations are caused by seasonal allergens whose pollination do not overlap with the study period.
6. Women of childbearing potential must have a negative urine pregnancy test at Screening visit/Visit 0
7. Women of childbearing potential must agree to use an appropriate contraception method during the study if they are sexually active

Exclusion Criteria:

1. Stable and continued use of medication for allergic pathology during 2 weeks prior to inclusion.
2. Patients sensitised to other perennial allergens clinically relevant and with specific IgE levels greater or equal to class 2 CAP/PHADIA.
3. Patients who received immunotherapy in the previous 5 years for DPT or for any allergen with cross reactivity or patients that are currently receiving immunotherapy for any allergen.
4. Patients with severe asthma or FEV1 minor than 70% or asthma requiring inhaled or systemic corticoid treatment at the time of study entry or within 8 weeks prior to treatment initiation.
5. Patients with: immunological, cardiac, renal or hepatic illnesses or any other medical condition that the investigator deems relevant so as to interfere with the study.
6. Patients with a previous history of anaphylaxis
7. Patients with chronic urticaria
8. Patients with unstable angina
9. Patients with uncontrolled hypertension
10. Patients with clinically significant arrythmias
11. Patients with neoplasia
12. Patients with clinically relevant malformations of the upper respiratory tract.
13. Other chronic or immunological disease that could interfere with the assessment of the investigational product or that could generate any additional risk for the patients
14. Patients who have participated in another clinical trial within 3 month prior to enrolment.
15. Patients under treatment with tricyclic antidepressives, psychotropics beta-blockers, or Angiotensin Converting Enzyme Inhibitors (ACEI)
16. Female patients who are pregnant or breast-feeding or women of childbearing potential that do not agree to use an appropriate contraception method during the study if they are sexually active, if they have not been surgically sterilised or present any other incapacity to bear
17. Patient who does not attend the visits
18. Patient's lack of collaboration or refusal to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mª Dolores Hernández, MD, Principal Investigator — Hospital Universitario La Fe; Ignacio Antépara, MD, Principal Investigator — Hospital de Basurto
Locations (2):
- Spain (2):
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital La Fe, Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A Active; Group A Placebo: 6 administrations and 5 weeks duration
  1. Vial 2: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals
  2. Vial 3: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals.
  subcutaneous immunotherapy with DPT extract: Increasing doses of subcutaneous immunotherapy in three different scales up to the maximum dose of 500 TSU (Treatment Standardized Units)
- Group B Active; Group B Placebo: 8 administrations and 7 weeks duration
  1. Vial 1: 0.2 ml at 1 week intervals
  2. Vial 2: 0.1 ml, 0.2 ml, 0.4 ml at 1 week intervals
  3. Vial 3: 0.1 ml, 0.2 ml, 0.4 ml and 0.5 ml at 1 week intervals
  subcutaneous immunotherapy with DPT extract: Increasing doses of subcutaneous immunotherapy in three different scales up to the maximum dose of 500 TSU (Treatment Standardized Units)
- Group C Active: 8 administrations, 2 administrations in the same day. 1 week interval between 2 doses, during 3 weeks.
  1. Week 1: vial 2 - 2 administrations of 0.1 ml with 30 minute interval
  2. Week 2: vial 2 - 0.2 ml and 0.3 ml with 30 minute interval
  3. Week 3: vial 3 - 2 doses of 0.1 ml with 30 minute interval
  4. Week 4: vial 3 - 0.2 ml and 0.3 ml with 30 minute interval
  subcutaneous immunotherapy with DPT extract: Increasing doses of subcutaneous immunotherapy in three different scales up to the maximum dose of 500 TSU (Treatment Standardized Units)
- Group C Placebo: 8 administrations, 2 administrations in the same day. 1 week interval between 2 doses, during 3 weeks.
  1. Week 1: vial 2 - 2 administrations of 0.1 ml with 30 minute interval
  2. Week 2: vial 2 - 0.2 ml and 0.3 ml with 30 minute interval
  3. Week 3: vial 3 - 2 dose of 0.1 ml with 30 minute interval
  4. Week 4: vial 3 - 0.2 ml and 0.3 ml with 30 minute interval
  subcutaneous immunotherapy with DPT extract: Increasing doses of subcutaneous immunotherapy in three different scales up to the maximum dose of 500 TSU (Treatment Standardized Units)
Period: Overall Study
Arm/Group | Group A Active | Group A Placebo | Group B Active | Group B Placebo | Group C Active | Group C Placebo
Started | 12 | 4 | 12 | 4 | 12 | 4
Completed | 11 | 4 | 9 | 4 | 6 | 4
Not Completed | 1 | 0 | 3 | 0 | 6 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0 | 3 | 0
Not completed — Concomitant disease | 0 | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A Active: 6 administrations and 5 weeks duration
  1. Vial 2: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals
  2. Vial 3: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals.
  subcutaneous immunotherapy with DPT extract: Increasing doses of subcutaneous immunotherapy in three different scales up to the maximum dose of 500 TSU (Treatment Standardized Units) or placebo
- Group B Active: 8 administrations and 7 weeks duration
  1. Vial 1: 0.2 ml at 1 week intervals
  2. Vial 2: 0.1 ml, 0.2 ml, 0.4 ml at 1 week intervals
  3. Vial 3: 0.1 ml, 0.2 ml, 0.4 ml and 0.5 ml at 1 week intervals
  subcutaneous immunotherapy with DPT extract: Increasing doses of subcutaneous immunotherapy in three different scales up to the maximum dose of 500 TSU (Treatment Standardized Units) or placebo
- Group C Active: 8 administrations, 2 administrations in the same day. 1 week interval between 2 doses, during 3 weeks.
  1. Week 1: vial 2 - 2 administrations of 0.1 ml with 30 minute interval
  2. Week 2: vial 2 - 0.2 ml and 0.3 ml with 30 minute interval
  3. Week 3: vial 3 - 2 doses of 0.1 ml with 30 minute interval
  4. Week 4: vial 3 - 0.2 ml and 0.3 ml with 30 minute interval
  subcutaneous immunotherapy with DPT extract: Increasing doses of subcutaneous immunotherapy in three different scales up to the maximum dose of 500 TSU (Treatment Standardized Units) or placebo
- Group A Placebo: 6 administrations and 5 weeks duration
  1. Vial 2: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals
  2. Vial 3: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals.
  Subcutaneous depot placebo
- Group B Placebo: 8 administrations and 7 weeks duration
  1. Vial 1: 0.2 ml at 1 week intervals
  2. Vial 2: 0.1 ml, 0.2 ml, 0.4 ml at 1 week intervals
  3. Vial 3: 0.1 ml, 0.2 ml, 0.4 ml and 0.5 ml at 1 week intervals
  subcutaneous depot placebo
- Group C Placebo: 8 administrations, 2 administrations in the same day. 1 week interval between 2 doses, during 3 weeks.
  1. Week 1: vial 2 - 2 administrations of 0.1 ml with 30 minute interval
  2. Week 2: vial 2 - 0.2 ml and 0.3 ml with 30 minute interval
  3. Week 3: vial 3 - 2 doses of 0.1 ml with 30 minute interval
  4. Week 4: vial 3 - 0.2 ml and 0.3 ml with 30 minute interval
  subcutaneous depot placebo
- Total: Total of all reporting groups
Arm/Group | Group A Active | Group B Active | Group C Active | Group A Placebo | Group B Placebo | Group C Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 4 | 4 | 4 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.66 (8.93) | 30.88 (9.77) | 31.80 (8.85) | 33.93 (9.49) | 33.93 (9.49) | 33.93 (9.49) | 32.68 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 7 | 3 | 2 | 1 | 24
  Male | 5 | 8 | 5 | 1 | 2 | 3 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number and Seriousness of Both Local and Systemic Adverse Reactions
Description: The primary end points were the number of ARs and the severity of local and systemic ARs (SARs) to SCIT administration. Proportions were compared between study arms. The tolerability of SCIT was evaluated by early and late local reactions (i.e., local swelling and redness) and systemic reactions after each injection (any symptoms from organs distant from the location of the injection). Reactions were classified depending on the severity and onset of the reaction, according to the EAACI classification (Alvarez-Cuesta 2006).
Time Frame: From informed consent signature (V0) until the end of patient participation in the study (depending on the treatment assigned between 4 and 8 weeks )
Measure: Number; unit: adverse reactions number
Arm/Group | Group A Active | Group B Active | Group C Active | Group A Placebo | Group B Placebo | Group C Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 4 | 4 | 4
adverse reactions number
  Local adverse reactions number | 2 | 1 | 0 | 1 | 1 | 0
  Systemic adverse reactions number | 4 | 6 | 4 | 0 | 1 | 1

2. Secondary Outcome: Immunoglobulin Levels (IgE Specific) Active Versus Placebo
Description: Changes on immunoglobulin level determinations (specific IgE, IgG and IgG4) from basal visit to final visit and changes in mean wheal area in prick test dose response from basal visit to final visit, active versus placebo.
Time Frame: Before (V0) and after treatment (depending on the treatment assigned between 4 and 8 weeks)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A Active | Group A Placebo | Group B Active | Group B Placebo | Group C Active | Group C Placebo
Number analyzed (Participants) | 11 | 4 | 9 | 4 | 6 | 4
ng/mL | 0.0750 (0.393) | -0.0055 (0.013) | 0.1709 (0.274) | -0.1445 (0.639) | -0.0398 (0.507) | 0.0395 (0.039)

3. Secondary Outcome: Immunoglobulin Levels (IgG Total) Active Versus Placebo
Description: Changes on immunoglobulin level determinations (IgG) from basal visit to final visit and changes in mean wheal area in prick test dose response from basal visit to final visit, active versus placebo.
Time Frame: Before (V0) and after treatment (depending on the treatment assigned between 4 and 8 weeks)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A Active | Group A Placebo | Group B Active | Group B Placebo | Group C Active | Group C Placebo
Number analyzed (Participants) | 11 | 4 | 9 | 4 | 6 | 4
ng/mL | -0.8813 (0.484) | -0.0405 (0.097) | -0.9589 (0.536) | -0.0953 (0.137) | -0.4918 (0.389) | -0.0425 (0.090)

4. Secondary Outcome: Immunoglobulin Levels (IgG 4) Active Versus Placebo
Description: Changes on immunoglobulin level determinations (IgG4) from basal visit to final visit and changes in mean wheal area in prick test dose response from basal visit to final visit, active versus placebo.
Time Frame: Before (V0) and after treatment (depending on the treatment assigned between 4 and 8 weeks)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A Active | Group A Placebo | Group B Active | Group B Placebo | Group C Active | Group C Placebo
Number analyzed (Participants) | 11 | 4 | 9 | 4 | 6 | 4
ng/mL | -1.0878 (0.770) | 0.0838 (0.518) | -1.2885 (0.844) | 0.0770 (0.162) | -0.8243 (0.663) | 0.0580 (0.039)

ADVERSE EVENTS:
Arm/Group | Group A Active | Group B Active | Group C Active | Group A Placebo | Group B Placebo | Group C Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/12 | 3/12 | 3/12 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 12/12 | 11/12 | 8/12 | 1/4 | 2/4 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Active (N=12) | Group B Active (N=12) | Group C Active (N=12) | Group A Placebo (N=4) | Group B Placebo (N=4) | Group C Placebo (N=4)
Otitis (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | NA | NA | NA
pyrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | NA | NA | NA
Facial edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | NA | NA | NA
urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | NA | NA | NA
Edema in upper extremities (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | NA | NA | NA
broncoconstriction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | NA | NA | NA
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA
allergic rhinoconjunctivitis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Active (N=12) | Group B Active (N=12) | Group C Active (N=12) | Group A Placebo (N=4) | Group B Placebo (N=4) | Group C Placebo (N=4)
cephalea (Nervous system disorders) | 3 (7) | 5 (12) | 4 (7) | 0 (0) | 1 (1) | 0 (0)
Cold (Infections and infestations) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
alterations injection site (General disorders) | 5 (12) | 7 (16) | 5 (20) | 1 (1) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No